CLINICAL TRIAL: NCT03326895
Title: A Prospective, Multi-Center Evaluation of the ECHELON CIRCULAR Powered Stapler in Left-Sided Colorectal Anastomoses
Acronym: EPMCS-CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESC-16-002
Record Dates: First submitted 2017-10-09; First posted 2017-10-31 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Left-sided Colon Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Group 1 (Experimental): Powered circular stapler used to complete anastomosis of colon
  Interventions: Device: Left-sided colon resection

INTERVENTIONS:
Device: Left-sided colon resection — Left-sided colon resection with powered stapler

SUMMARY:
This prospective clinical study will evaluate the intra-operative performance of the powered circular stapler used in left colectomy procedures in a post-market setting.

DETAILED DESCRIPTION:
Surgical staplers have been utilized in colorectal procedures since the early 20th century, with intraluminal staplers used to create the anastomosis since 1979. Successful utilization of these devices, whether in open or laparoscopic procedures, requires extensive training and experience. Even with experience, device issues such as stapler misfire, incomplete firing, low surgeon satisfaction, etc., may occur. In a retrospective study of 349 colorectal resections, 67 (19%) procedures had some type of technical error. The most frequently reported issues from the analysis were positive leak tests, difficulty placing or removing the stapler, and inadequate donuts. Surgeons may also experience psychological or physical stress during procedures due to complications, workload, or other factors.

Patients scheduled to undergo a left-sided colon resection, and who meet study entry criteria, may be enrolled. Investigators will perform each procedure using the powered circular stapler according to the instructions for use (IFU). There will be no blinding or planned-interim analysis. Procedures may be performed open or via minimally invasive surgery (MIS) according to institutional standard-of-care (SOC). Use of a hand port and robotic assistance are permissible providing the powered circular stapler is used to create the anastomosis. Conversion from laparoscopic to open surgery is permissible under the protocol at the surgeon's discretion for the patient's safety.

The final scheduled study visit will occur 28 days post-procedure (routinely scheduled follow-up with surgeon). Follow-up by phone is permissible when an on-site visit is not planned or is more than six weeks post-operative.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for colectomy with left-sided anastomosis peformed with a circular stapler;
2. Willing to give consent and comply with all study-related evaluations; and
3. At least 18 years of age.

Exclusion Criteria:

1. Enrollment in a concurrent clinical study;
2. Pregnancy;
3. Physical or psychological condition which would impair study participation;
4. Emergency surgery;
5. ASA Class ≥ IV;
6. The subject is judged unsuitable for study participation by the Investigator; or
7. Unable or unwilling to provide follow-up information 8, Undergoing multiple intraoperative synchronous colon resections;

9. Anastomosis not distal from splenic flexure of the colon 10. Anastomosis of the colon not attempted 11. Subjects with any intraoperative findings identified by the surgeon that would preclude attempting an anastomosis with a circular stapler.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Herzig, MD, Principal Investigator — Oregon Health and Science University
Locations (12):
- United States (6):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Colon & Rectal Clinic of Orlando, Orlando, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Spectrum Health System, Grand Rapids, Michigan
  - Mt. Sinai Hospital / Mt. Sinai School of Medicine, New York, New York
  - Oregon Health & Science University, Portland, Oregon
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Schon Klinik Neustadt, Neustadt, Germany
- Hospital Universitario Virgen Rocio, Seville, Spain
- United Kingdom (3):
  - University Hospitals Birmingham NHS, Birmingham
  - St Jame's University Hospital, Leeds
  - St. Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Primary endpoint

REFERENCES:
- [Result] Herzig DO, Ogilvie JW, Chudzinski A, Ferrara A, Ashraf SQ, Jimenez-Rodriguez RM, Van der Speeten K, Kinross J, Schimmelpenning H, Sagar PM, Cannon JA, Schwiers ML, Singleton DW, Waggoner JR, Fryrear R 2nd, Sylla P. Assessment of a circular powered stapler for creation of anastomosis in left-sided colorectal surgery: A prospective cohort study. Int J Surg. 2020 Dec;84:140-146. doi: 10.1016/j.ijsu.2020.11.001. Epub 2020 Nov 8. PMID 33176211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects who underwent surgery and had an anastomosis attempted with the ECHELON CIRCULAR Powered stapler were included in performance and safety analyses.
Groups:
- ECHELON CIRCULAR Powered Stapler: Use of the ECHELON CIRCULAR Powered Stapler
Period: Overall Study
Arm/Group | ECHELON CIRCULAR Powered Stapler
Started (168) | 168
Completed (168) | 168
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ECHELON CIRCULAR Powered Stapler
Number analyzed (Participants) | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 152
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 149
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stapler Performance Issues
Description: A stapler performance issue is defined as a failure of the ECHELON CIRCULAR Powered Stapler to perform per its instructions for use. This includes but is not limited to difficulty placing or removing the stapler, stapler misfire/failure of the device to fully fire, staple line defects, incomplete or thin donuts, tissue damage, positive intraoperative leak test, detached components, unformed staples, or any other device failure.
Time Frame: Intraoperative
Population: Number of subjects with at least performance issue.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ECHELON CIRCULAR Powered Stapler
Number analyzed (Participants) | 168
Percentage of subjects | 11.9 [7.4 to 17.8]

2. Secondary Outcome: SURG-TLX Questionnaire
Description: The Surgery Task Load index (SURG-TLX) questionnaire was completed by the participating surgeon following each procedure. The questionnaire was used to provide an assessment of surgical stress (surgeon) associated with the procedure (defined as the creation of the anastomosis).
  There are six specific components (mental, physical, temporal, task, situational, and distractions) that are used for evaluating the surgeon experience after each surgery is performed. Each component is scored on a 0 to 100 scale with lower scores representing a "low" response on that component and higher scores indicating a "high" response on that component. An overall score is also calculated as the average of the six components for each procedure.
Time Frame: Collected postoperative for intraoperative stress
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | ECHELON CIRCULAR Powered Stapler
Number analyzed (Participants) | 168
Scores on a Scale
  Overall Score | 38.0 (21.60)
  Mental Demands (How mentally fatiguing was the procedure?) | 44.9 (27.8)
  Physical Demands (How physically fatiguing was the procedure?) | 37.9 (26.5)
  Temporal Demands (How hurried or rushed was the pace of the procedure?) | 30.3 (22.6)
  Task Complexity (How complex was the procedure?) | 50.3 (28.6)
  Situational Stress (How anxious did you feel while performing the procedure?) | 38.6 (27.3)
  Distractions (How distracting was the operating environment?) | 26.5 (21.0)

ADVERSE EVENTS:
Time Frame: 4 Weeks Post Procedure
Arm/Group | ECHELON CIRCULAR Powered Stapler
All-Cause Mortality (participants affected / at risk) | 0/168
Serious Adverse Events (participants affected / at risk) | 13/168
Other Adverse Events (participants affected / at risk) | 32/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ECHELON CIRCULAR Powered Stapler (N=168)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 3
Anastomotic Leak (Injury, poisoning and procedural complications) | 2
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 1
Incision Site Pain (Injury, poisoning and procedural complications) | 1
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 1
Post-operative Ileus (Injury, poisoning and procedural complications) | 1
Stoma Complication (Injury, poisoning and procedural complications) | 1
Stoma Site Erythema (Injury, poisoning and procedural complications) | 1
Pelvic Abscess (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 1
C-reactive Protein Increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ECHELON CIRCULAR Powered Stapler (N=168)
Abdominal Pain (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Procedural Pain (Injury, poisoning and procedural complications) | 5
Acute Kidney Injury (Renal and urinary disorders) | 4
Urinary Retention (Renal and urinary disorders) | 3
Oxygen Saturation Decreased (Investigations) | 3
Pyrexia (General disorders) | 4
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT03326895/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT03326895/SAP_001.pdf